CLINICAL TRIAL: NCT01063205
Title: N-AcetylCysteine as a Potential Treatment of Methamphetamine Dependence
Brief Title: NAC as a Potential Treatment for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas Newton, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-24927; DPMC (Other: NIDA); R21DA024756 (NIH)
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Methamphetamine Abuse; Methamphetamine Dependence; Substance Abuse
Keywords: Methamphetamine; NAC; N-acetylcysteine
MeSH Terms: conditions — Substance-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- N-Acetylcysteine (NAC) 1800 mg (Active Comparator)
  Interventions: Drug: N-acetylcysteine
- N-Acetylcysteine (NAC) 3600 mg (Active Comparator)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: Placebo — Placebo administration will be started on day 2 and stopped on day 5. Methylsulonylmethane (MSM) will serve as a placebo for MA.
  Other Names: Methylsulonylmethane (MSM)
  Arms: Placebo
Drug: N-acetylcysteine — Study medication (NAC 1800 mg) will be started on day 2 and stopped on day 5.
  Other Names: NAC
  Arms: N-Acetylcysteine (NAC) 1800 mg
Drug: N-acetylcysteine — Study medication (NAC 3600 mg) will be started on day 2 and stopped on day 5.
  Other Names: NAC
  Arms: N-Acetylcysteine (NAC) 3600 mg

SUMMARY:
The purpose of this study is to determine the effects of treatment with NAC, compared to treatment with placebo, on cue- and methamphetamine (MA)-induced craving and MA subjective effects in non-treatment-seeking MA-dependent human volunteers. We also aim to determine the effects of treatment with NAC, compared to treatment with placebo, on the reinforcing effects of MA by measuring MA self-administration in non-treatment-seeking MA-dependent human volunteers.

DETAILED DESCRIPTION:
N-acetyl-l-cysteine (NAC) treatment is associated with reduced susceptibility to reinstatement of cocaine seeking behavior in rats (Baker et al 2002) and with reduced cue-induced craving in cocaine-dependent human volunteers (LaRowe et al 2006). We propose these aims to evaluate the potential of NAC as a treatment for methamphetamine (MA) dependence: Specific Aim 1: To determine the effects of treatment with NAC(placebo, 1800 and 3600mg daily), compared to treatment with placebo, on cue- and MA-induced craving and MA subjective effects in non-treatment-seeking MA-dependent human volunteers. We hypothesize that treatment with NAC will reduce craving for MA reported following exposure to MA cues and will reduce craving and MA subjective effects reported following non-contingent administration of MA (0mg,9mg, and 30 mg, IV). Specific Aim 2: To determine the effects of treatment with NAC (placebo, 1800 and 3600mg daily), compared to treatment with placebo, on the reinforcing effects of MA by measuring MA self-administration in non-treatment-seeking MA-dependent human volunteers. We hypothesize that treatment with NAC will reduce the number of choices made for MA during choice sessions.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking non-treatment-seeking volunteers.
* Be between 18-55 years of age.
* Meet DSM-IV TR criteria for MA dependence.
* Have a self-reported history of using MA by the smoked route.
* Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 85-150mm Hg systolic and 45-90mm Hg diastolic.
* Have a breathalyzer test indicating an undetectable blood alcohol level upon admission.
* Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal.
* Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias.
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator. Adult ADHD is allowable, as long as symptoms do not interfere with participation.

Exclusion Criteria:

* Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure.
* Have neurological or psychiatric disorders, such as: a. episode of major depression within the past 2 years as assessed by MINI; b. lifetime history of schizophrenia, other psychotic illness, or bipolar illness as assessed by MINI; c. current organic brain disease or dementia assessed by clinical interview; d. history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; e. history of suicide attempts within the past year and/or current suicidal ideation/plan. f. history of psychosis occurring in the absence of current MA use.
* Meet DSM-IV criteria for abuse or dependence on alcohol or other drugs, except for nicotine.
* Meet DSM-IV criteria for dependence on marijuana.
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI.
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
* Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication.
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation.
* Currently use alpha or beta agonists, theophylline, or other sympathomimetics.
* Have any other illness, condition, or use of medications, which in the opinion of the P.I. and/or the admitting physician would preclude safe and/or successful completion of the study.
* Have sulfur allergy.

Criteria for Discontinuation Following Initiation:

Participants will be discharged if they have a positive urine toxicology or breath test indicating illicit use of drugs while on the Research Commons, if they do not comply with study procedures, or if they do not tolerate MA. MA will not be administered if participants do not continue to meet inclusion criteria listed above or if the study physician believes there may be any reason to withhold MA.

Rationale for Subject Selection Criteria:

Participants are required to have used MA by the intravenous route in order to avoid exposing participants to new routes of administration. Participants with asthma or who take medications for asthma are excluded due to potential adverse interactions between treatment medications and MA. Participants who use alcohol heavily are excluded due to the potential of withdrawal symptoms in the hospital. Participants with active HIV disease are excluded to avoid potentially exacerbating their underlying illness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The effects of treatment with NAC (placebo, 1800 and 3600 mg daily), compared to treatment with placebo, on cue- and MA-induced craving and subjective effects in MA-dependent human volunteers.
  On days 3-5, participants will take part in active cues and neutral cues. On days 4 and 5, they will make choices to receive MA/placebo in a self-administration paradigm. Participants will also rate craving, desire, and would take MA if available on a 0-100 mm visual analogue scale.

SECONDARY OUTCOMES:
The effects of treatment with NAC (placebo, 1800 and 3600 mg daily), compared to treatment with placebo, on the reinforcing effects of MA by measuring MA self-administration in MA-dependent human volunteers.
  On days 4 and 5, participants will make choices to receive MA/placebo in a self-administration paradigm. Any alterations in the reinforcing effects of MA associated with NAC treatment will be evident as changes in the number of choices made for MA.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States